CLINICAL TRIAL: NCT07290985
Title: AACR Adaptive Biomarker-Driven Organ Preservation Trial In Gastroesophageal Adenocarcinomas (AACR-ADOPT-GEA)
Brief Title: AACR Adaptive Biomarker-Driven Organ Preservation Trial in Gastroesophageal Adenocarcinomas
Acronym: AACR-ADOPT-GEA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: American Association for Cancer Research (Other)
Collaborators: Jazz Pharmaceuticals (Industry); BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AACR-ADOPT-GEA
Record Dates: First submitted 2025-11-17; First posted 2025-12-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gastroesophageal Adenocarcinoma
MeSH Terms: interventions — tislelizumab; Leucovorin; Oxaliplatin; Fluorouracil; zanidatamab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zanidatamab + Tislelizumab (HER2) Sub-Study (Experimental): Patients will receive zanidatamab on Day 1 of each 14-day cycle, followed by tislelizumab and mFOLFOX6 chemotherapy: leucovorin (Day 1), oxaliplatin (Day 1), and 5-FU as a 48-hour continuous intravenous infusion (Days 1-2). Up to 8 preoperative cycles will be given, followed by surgery or organ preservation if a complete response is achieved. Post-surgery or organ preservation, zanidatamab + tislelizumab will continue every 2 weeks for up to 1 year of perioperative therapy.
  Interventions: Drug: Tislelizumab; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Fluorouracil; Drug: Zanidatamab

INTERVENTIONS:
Drug: Tislelizumab — 150 mg every 2 weeks for 4 months pre-operatively and up to 8 months post-operatively
Drug: Leucovorin — 400 mg/m² every 2 weeks for 4 months pre-operatively and up to 8 months post-operatively
Drug: Oxaliplatin — 85 mg/m² every 2 weeks for 4 months pre-operatively and up to 8 months post-operatively
Drug: Fluorouracil — 2,400 mg/m² every 2 weeks for 4 months pre-operatively and up to 8 months post-operatively
Drug: Zanidatamab — 1,200 mg for patients weighing less than 70 kg and 1,600 mg for patients weighing 70 kg or more every 2 weeks for 4 months pre-operatively and up to 8 months post-operatively

SUMMARY:
This study will test a new personalized treatment approach for patients with stomach or esophageal cancer. It will take place in two stages and aims to find the best combination of chemotherapy, immunotherapy, and targeted drugs based on each patient's tumor biomarkers.

Upon enrollment onto the study, patients will consent to tumor biomarker testing and may receive one cycle of standard chemotherapy while awaiting results. Those with a matching biomarker will join the corresponding treatment group that combines chemotherapy, an immune checkpoint inhibitor, and/or a targeted therapy. In Stage I of the study, treatment lasts about four months before surgery, followed by an additional eight months of therapy for a total of one year.

The most effective treatments from Stage I will be studied further in Stage II of the study to see whether some patients can safely avoid surgery. Those patients enrolled during Stage II will receive four months of the same combination treatment (chemotherapy, an immune checkpoint inhibitor, and/or a targeted therapy) but may be eligible to skip surgery if their cancer completely disappears after pre-surgery therapy. All patients will then receive an additional eight months of therapy and those who skipped surgery will be closely monitored with scans and endoscopies.

DETAILED DESCRIPTION:
This is a two-stage, prospective, multi-center, perioperative, biomarker-driven, open-label study. The trial design consists of a screening phase (Stage I) and a testing phase (Stage II).

Stage I:

Eligible patients will provide screening consent and research tissue for biomarker assessment. While awaiting results, they may receive one cycle of FLOT or mFOLFOX6. Once a biomarker included in the study platform is identified, patients will sign a second consent and be assigned to the corresponding subgroup. They will continue treatment with the chemotherapy backbone (mFOLFOX6) plus an immune checkpoint inhibitor and a biomarker-targeted agent. Patients who began on FLOT will switch to mFOLFOX6 once a targeted agent is added. If no actionable biomarker is detected, patients will continue standard-of-care therapy off-study. Patients receiving the chemotherapy + immune checkpoint inhibitor + targeted agent combination will complete 4 months of preoperative therapy, followed by surgery and postoperative therapy for a total treatment duration of up to one year. Once 24 patients in a given biomarker subgroup have undergone surgery, continuation to Stage II will depend on meeting predefined efficacy thresholds. Only regimens demonstrating sufficient efficacy will advance.

Stage II:

Effective therapies identified in Stage I will be further evaluated to establish predictive markers of pathological complete response (pathCR) and identify patients who may safely avoid surgery. Patients will provide tissue for central biomarker testing and may receive a chemotherapy cycle while awaiting results. Once assigned to an eligible biomarker subgroup, they will receive mFOLFOX6 + immune checkpoint inhibitor plus the targeted agent for 4 months. Response will be assessed through clinical, endoscopic, and radiologic evaluation. Patients showing no residual disease after preoperative therapy will forgo surgery and continue maintenance therapy (immune checkpoint inhibitor plus the targeted agent) for an additional 8 months with regular surveillance. Those with residual disease will proceed to surgery, followed by postoperative therapy and follow-up for up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, resectable adenocarcinoma of the stomach, esophagus, or gastroesophageal junction (Stage II or higher, T2N0 with high-risk features).
* Complete surgical resection deemed achievable by multidisciplinary evaluation.
* Willingness to undergo tumor biopsies for biomarker analysis (HER2, FGFR2b, PD-L1, MSI) at screening, progression, or pre/post- surgery.
* Life expectancy ≥ 24 weeks. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
* Adequate organ function:

  * Hematologic: absolute neutrophil count (ANC) ≥1.5 ×10⁹/L, platelets ≥100 ×10⁹/L, hemoglobin ≥ 8 g/dL
  * Hepatic: aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) ≤2.5 × ULN, total bilirubin ≤1.5 × upper limit of normal (ULN) (≤2.5 × ULN for Gilbert's)
  * Renal: creatinine ≤1.5 × ULN or creatinine clearance ≥50 mL/min/1.73 m²
* Willingness for blood samples to be drawn for research purposes.
* Baseline dihydropyrimidine dehydrogenase (DPD) testing per local guidelines; dosing of 5-FU adjusted for deficiency.
* Use of two effective contraception methods for women of childbearing potential and men during and 4 months after study; pregnant or breastfeeding women excluded.
* Must have the ability to understand and the willingness to sign a written informed consent document.
* Willingness and able to comply with the protocol for the duration of the study, including attending scheduled visits, examinations, the screening procedure, and having their tumor and blood molecularly characterized.
* Understands they must meet all Inclusion and Exclusion criteria in the sub-protocol for the treatment for which they will be later assigned

Additional inclusion criteria for all sub-studies:

• FFPE tumor sample tested at a central laboratory confirming PD-L1 Tumor Area Positivity (TAP) score ≥1%.

Additional inclusion criteria specific to HER2 sub-study:

* Histologically confirmed diagnosis of resectable (i.e., radical surgery eligible), HER2-positive (defined as 3+ HER2 expression by IHC or 2+ HER2 expression by immunohistochemistry (IHC) with in situ hybridization (ISH)-positivity per central assessment) adenocarcinoma of the stomach or esophagus, including the gastroesophageal junction.
* Formalin-fixed, paraffin-embedded (FFPE) tumor sample tested at a central laboratory confirming HER2-positive status.
* Left ventricular ejection fraction (LVEF) ≥50% as determined by either echocardiogram or multiple gated acquisition scan (MUGA).

Exclusion criteria:

* Unresectable disease, peritoneal dissemination, and/or positive cytology on laparoscopy.
* Peripheral neuropathy ≥ Grade 2.
* Active infection.
* Chronic growth factor support for white blood cells or granulocytes.
* Concurrent anti-cancer therapy (exceptions: supportive care medications ≥1 month prior, low molecular weight heparin, prior adjuvant hormonal therapy >3 years, palliative radiation

  ≤14 days prior).
* Local/systemic therapy for current gastroesophageal diagnosis (except one FLOX/ mFOLFOX6 dose during screening).
* Significant medical conditions compromising safety or protocol compliance.
* Preexisting cardiac conditions.
* Stroke, transient ischemic attack (TIA), or myocardial infarction within 6 months.
* Prior FGFR-targeted therapy.
* Prior HER2-targeted therapy (except >5 years prior for breast cancer).
* Prior checkpoint inhibitor therapy (anti-PD-1/PD- L1/PD-L2).
* Conditions preventing safe surgery/biopsy.
* Malabsorption syndrome or inability to swallow oral medication.
* Pregnant or nursing women
* History of stem cell or organ transplant.
* Major surgery within 14 days.
* Other malignancy within 3 years (exceptions: basal/squamous cell carcinoma, in situ malignancy, low-risk prostate cancer).
* Systemic corticosteroids >10 mg prednisone/ day or immunosuppressive therapy ≤14 days prior (exceptions: adrenal replacement, topical/ inhaled, short prophylactic courses).
* HIV with CD4 <350, active hepatitis B or C.
* Active or relapsing autoimmune disease (exceptions: controlled type I diabetes, hypothyroidism on replacement, controlled celiac disease, mild skin disease, other non- recurrent diseases).

Additional exclusion criteria for all sub-studies:

* History of hypersensitivity or contraindications to any active substance/active ingredient of any study medication, including chemotherapy components monoclonal antibodies, recombinant proteins, and/or any of the excipients listed in the ingredients of any drug formulation
* Poorly controlled seizures
* Clinically significant bleeding (CTCAE ≥ Grade 3) from the gastrointestinal (GI) tract within 4 weeks prior to enrollment.
* Administered a live vaccine ≤ 4 weeks prior to enrollment
* History of interstitial lung disease or non-infectious pneumonitis, or with severe dyspnea at rest or requiring supplementary oxygen therapy.
* Treated with another investigational product within 28 days of enrolment.

Exclusion criteria specific to HER2 sub-study:

* Total lifetime anthracycline load exceeding 360 mg/m² of doxorubicin or equivalent
* QTc Fridericia (QTcF) >470 ms. Note: For subjects with longer QTcF on initial electrocardiogram (ECG), follow-up ECG may be performed in triplicate to determine eligibility (e.g., after correction of electrolyte abnormalities, or discontinuation of QT-prolonging drugs).
* Ongoing Grade 2 or greater diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pathCR) Rate (Stage I). | At time of surgery.
  Proportion of patients achieving a pathCR in the surgical specimen after perioperative biomarker-directed systemic therapy.
Organ Preservation Rate (Stage II) | Up to 12 months post-treatment.
  Proportion of patients able to avoid surgery and preserve the affected organ due to biomarker-driven treatment response.

SECONDARY OUTCOMES:
Event-Free Survival (Stage I). | Up to 24 months post-treatment.
  : Time from initiation of treatment to the first documented disease progression, recurrence, or death from any cause.
Overall Survival (Stage I). | Up to 24 months post-treatment.
  Time from initiation of treatment to death from any cause.
Tumor Regression Grade. | At time of surgery (Stage I).
  Assessment of tumor response in surgical specimens using National Comprehensive Cancer Network (NCCN) guidelines.
Correlation between event-free survival and changes in circulating tumor DNA concentration. | Through study completion, an average of 3 years for Stage I and 6 years for Stage II.
  Correlation between event-free survival (defined as time from initiation of treatment to the first documented disease progression, recurrence, or death from any cause) and plasma ctDNA concentration (mean tumor molecules per milliliter) measured using a personalized, tumor-informed assay.
Correlation between overall survival and changes in circulating tumor DNA concentration. | Through study completion, an average of 3 years for Stage I and 6 years for Stage II.
  Correlation between overall survival (defined as time from initiation of treatment to death from any cause) and plasma ctDNA concentration (mean tumor molecules per milliliter) measured using a personalized, tumor-informed assay.
Correlation between tumor regression grade (TRG) and changes in circulating tumor DNA concentration. | Through study completion, an average of 3 years for Stage I and 6 years for Stage II.
  Correlation between tumor regression grade (TRG 1, 2, or 3 per NCCN guidelines) and plasma ctDNA concentration (mean tumor molecules per milliliter) measured using a personalized, tumor-informed assay.
Treatment-Related Toxicity and Tolerability (Stage I) | During treatment and up to 30 days post-treatment.
  Incidence and severity of adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) v6.0.

IPD SHARING:
Plan to Share IPD: No